CLINICAL TRIAL: NCT04434352
Title: Low Intensity Shockwave Therapy for Erectile Dysfunction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Ryan Smith, MD, Associate Professor of Urology, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-HSR# 190082
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Erectile Dysfunction; Erectile Dysfunction Following Radical Prostatectomy; Erectile Dysfunction Following Radiation Therapy; Erectile Dysfunction Due to General Medical Condition; Erectile Dysfunction Due to Arterial Insufficiency
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be randomized to either the treatment group or sham group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Baseline Erectile Dysfunction (Active Comparator): The first arm of the study will be those men with erectile dysfunction as defined by IIEF score. These men will either have PDE5i refractory or responsive erectile dysfunction. Subjects will receive either Sham treatment (no ultrasound energy delivered via a Sham probe) or LiSWT for erectile dysfunction. Follow up will occur at 1 month, 3 months, and 6 months following the end of treatment. Effectiveness will be measured by change in IIEF/SHIM score and EHS score. Each questionnaire is described in the trial description with a higher score indicating improved function.
  Interventions: Device: Storz Duolith Low-Intensity Shockwave Therapy
- Erectile Dysfunction-Penile Rehabilitation (Active Comparator): The second population of patients will be those who are planning to undergo treatment for prostate cancer. In a similar manner, men will be randomized to either the Sham or active treatment groups. Men will be treated prior to undergoing definitive treatment for prostate cancer to assess the effectiveness in LiSWT as a means of erectile preservation prior to prostate cancer treatment.
  Interventions: Device: Storz Duolith Low-Intensity Shockwave Therapy
- Erectile Dysfunction Post-Prostate Cancer Treatment (Active Comparator): The third population of patients will be those who have undergone treatment for prostate cancer. The investigators will compare IIEF scores and EHS scores in men who have undergone prostatectomy or radiation therapy. Again, there will be a sham and treatment group.
  Interventions: Device: Storz Duolith Low-Intensity Shockwave Therapy

INTERVENTIONS:
Device: Storz Duolith Low-Intensity Shockwave Therapy — A: Sham - the sham uses an attachment on the hand held probe that mimics the shockwave device, however it does not deliver any shockwaves. Sham will be delivered twice weekly for 3 weeks in the same manner as the LiSWT. The sham treatment will take about 20 minutes to complete.
  B: LiSWT delivered twice weekly for 3 weeks, comprising of 3000 shockwaves delivered to the distal penis (1000 shockwaves), base of penis (1000 shockwaves), and corporal bodies on the perineum (500 shockwaves to each crura). LiSWT is delivered into the penile tissue by a small hand held probe that produces low intensity shockwaves. A tranducer head is placed on the left and right sides of the penis. Treatment takes about 20 minutes to complete.
  Other Names: Sham

SUMMARY:
Low-intensity shockwave therapy (LiSWT) has been deemed "a safe and well-tolerated procedure but its efficacy for the treatment of ED is doubtful and deserves more investigation" by the European Society of Sexual Medicine. In a similar manner, the Sexual Medicine Society of North America and American Urological Association have put forth guideline statements recommending additional investigation of this treatment modality.2

The current clinical armamentarium only treats the symptoms of erectile dysfunction without improving upon the underlying pathophysiology. LiSWT has been used effectively in musculoskeletal disorders and cardiovascular applications. Animal studies have shown improvements in angiogenesis and stem cell recruitment in other systems (cardiac and musculoskeletal) using shockwave therapy. It has been used to treat erectile dysfunction since 2010 and is widely used in Europe and throughout the world. It is gaining widespread acceptance in the United States with a relative paucity of data in regards to its effectiveness.

While the majority of studies and meta-analyses show improvements in standardized erectile dysfunction questionnaires (IIEF/SHIM-Sexual Health Inventory in Men, International Index of Erectile Function-5) the durability remains unknown and many have lacked a sham-arm. In addition, many studies have failed to assess a population of men who have highly prevalent erectile dysfunction, those men undergoing prostate cancer treatment.

This is a prospective, randomized, single blind, sham-controlled clinical study aimed to evaluate the safety and efficacy of low-intensity shockwave therapy (LiSWT) on symptomatic ED patients in three distinct patient populations. LiSWT has shown the potential to improve baseline erectile function but requires further study, which is the aim of this investigation.

DETAILED DESCRIPTION:
It is estimated that about 1 in 10 adult males suffer from erectile dysfunction (ED) on a long-term basis. Oral therapies, including PDE5I, may be considered first-line therapies for the majority of patients with ED because of potential benefits and lack of invasiveness. This is a prospective, randomized, single-blind, sham-controlled clinical study aimed to evaluate the safety and efficacy of low-intensity shockwave therapy on symptomatic ED patients in three distinct patient populations.

The first arm of the study will be those men with erectile dysfunction as defined by IIEF score (International Index of Erectile Function-5). These men will either have PDE5i refractory or responsive erectile dysfunction. Subjects will receive either Sham treatment (no ultrasound energy delivered via a Sham probe) or LiSWT for erectile dysfunction. Follow up will occur at 1 month, 3 months, and 6 months following the end of treatment. Effectiveness will be measured by change in IIEF/SHIM (IIEF/SHIM-Sexual Health Inventory in Men, International Index of Erectile Function-5) score and EHS (Erection Hardness Score) score.

The Sexual Health Inventory in Men (also referred to as International Index of Erectile Function-5) is scored as follows:

22-25 No erectile dysfunction 17-21 Mild erectile dysfunction 12-16 Mild-to-moderate erectile dysfunction 8-11 Moderate erectile dysfunction 5-7 Severe erectile dysfunction

The patient responds to the following questions:

Instructions Each question has 5 possible responses. Circle the number that best describes your own situation.

Select only 1 answer for each question.

Over the past 6 months:

1. How do you rate your confidence that you could keep an erection? Very low (1), Low (2), Moderate (3), High (4), Very high (5)
2. When you had erections with sexual stimulation, how often were your erections hard enough for penetration (entering your partner)?

   Almost never or never (1), A few times (much less than half the time) (2), Sometimes (About half the time) (3), Most times (much more than half the time) (4), Almost always or always (5)
3. During sexual intercourse, how often were you able to maintain your erection after you had penetrated (entered) your partner?

   Almost never or never (1), A few times (much less than half the time) (2), Sometimes (About half the time) (3), Most times (much more than half the time) (4), Almost always or always (5)
4. During sexual intercourse, how difficult was it to maintain your erection to completion of intercourse?

   Extremely difficult (1), Very difficult (2), Difficult (3), Slightly difficult (4), Not difficult (5)
5. When you attempted sexual intercourse, how often was it satisfactory for you? Almost never or never (1), A few times (much less than half the time) (2), Sometimes (About half the time) (3), Most times (much more than half the time) (4), Almost always or always (5)

An increase or decrease from baseline indicates improving or worsening erectile function. The Erection Hardness score is another tool to evaluate erectile function and firmness. It is scored as follows:

0-Penis does not enlarge

1. Penis is larger, but not hard
2. Penis is hard, but not hard enough for penetration
3. Penis is hard enough for penetration, but not completely hard
4. Penis is completely hard and fully rigid

These patients will be randomized in a 1:1 ratio into either the Sham or active treatment groups in which a device called Duolith by Storz will be used to deliver shockwaves to the penile tissue. The Duolith device is FDA-approved for treatment of musculoskeletal disorders including plantar fasciitis but has more recently been investigated in erectile dysfunction in both the United States and abroad.

The Duolith device is used to deliver low intensity shockwaves to the penile tissue. LiSWT (Linear Shockwave Therapy) utilizes energy in the ultrasonic range. The focused energy, when applied to tissue, has been postulated to improve stem cell recruitment and promote angiogenesis. This has been demonstrated in animal modes.

The second population of patients will be those who are planning to undergo treatment for prostate cancer. In a similar manner, men will be randomized to either the Sham or active treatment groups. Men will be treated prior to undergoing definitive treatment for prostate cancer to assess the effectiveness in LiSWT as a means of erectile preservation prior to prostate cancer treatment.

The third population of patients will be those who have undergone treatment for prostate cancer. The investigators will compare IIEF scores and EHS scores in men who have undergone prostatectomy or radiation therapy. Again, there will be a sham and treatment group.

In addition to assessing the efficacy of LiSWT in these populations of men, the study aims also to substantiate the safety profile of the Duolith device. Safety is to be assessed by the frequency of side effects during treatment, as well as the occurrence of anticipated and unanticipated adverse events during and from treatment up to follow-ups. The average and standard deviation of all relevant variables, including demographic and baseline characteristics, primary and secondary outcomes will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be willing and able to provide informed consent.
* The patient is a male between >30 and <80 years of age.
* PDE5i responsive or non-responsive. If on PDE5i patient will discontinue medication for 2 weeks before baseline IIEF.
* Baseline IIEF-EF score ≥ 8 and ≤21. If taking PDE5i, stop medication for at least 4 weeks before baseline IIEF.
* Testosterone level > 300 ng/dL. This includes patients on therapeutic testosterone therapy.
* If diabetic, HgbA1C level ≤ 7.5% within 3 months prior to enrollment.
* Men who have undergone radical prostatectomy ≥ 12 months ago
* Men who have undergone radiation therapy, either brachytherapy or external bean therapy ≥ 12 months ago

Exclusion Criteria:

* History of extensive pelvic surgery ever.
* Past radiation therapy of the pelvic region within 12 months prior to enrollment.
* Recovering from any non-prostate related cancer within 12 months prior to enrollment.
* Neurological disease which affects erectile function at the discretion of the investigator.
* Anatomical malformation of the penis, including Peyronie's disease.
* Testosterone level <300 within 3 month prior to enrollment.
* HgbA1C level > 7.5% within 3 month prior to enrollment.
* History of spinal cord injury.
* Recovering from any non-prostate cancer malignancy within 12 months prior to enrollment.

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 338 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-01-09 (Estimated)

PRIMARY OUTCOMES:
Change in IIEF/SHIM score (International Index of Erectile-Function-5, Sexual Health Inventory in Men) Score at 1 month post-treatment | 1 month
  The primary outcome will be change in (International Index of Erectile-Function-5, Sexual Health Inventory in Men) score from baseline (pre-treatment) to 1 month after the end of treatment. The IIEF/SHIM score is a validated instrument to assess erectile function.
  Over the past 6 months:
  1. How do you rate your confidence that you could keep an erection?
  2. When you had erections with sexual stimulation, how often were your erections hard enough for penetration (entering your partner)?
  3. During sexual intercourse, how often were you able to maintain your erection after you had penetrated (entered) your partner?
  4. During sexual intercourse, how difficult was it to maintain your erection to completion of intercourse?
  5. When you attempted sexual intercourse, how often was it satisfactory for you? Each item is scored 1-5, with a higher number indicating better rigidity.

SECONDARY OUTCOMES:
Changes in (International Index of Erectile-Function-5, Sexual Health Inventory in Men) at 3 and 6 months post-treatment | 3 and 6 months
  Changes in SHIM score (Sexual Health Inventory in Men) score at 3 and 6 months post-treatment.
  • The IIEF classifies men into groups of no erectile dysfunction, mild, mild to moderate, moderate and severe erectile dysfunction. Changes in the classifications will be compared between arms at 1, 3, and 6 months post-treatment.
Adverse Event Rates | 1, 3 and 6 months
  Adverse Events including bruising and pain.
Change in Erection Hardness Score at 1, 3, and 6 months | 1, 3, and 6 months
  Change in Erection Hardness Score
  The Erection Hardness score is another tool to evaluate erectile function and firmness. It is scored as follows:
  0-Penis does not enlarge
  1. Penis is larger, but not hard
  2. Penis is hard, but not hard enough for penetration
  3. Penis is hard enough for penetration, but not completely hard
  4. Penis is completely hard and fully rigid
  A higher score indicates a higher degree of erectile rigidity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lange M, Charles D, Kazeem A, Jones M, Sun F, Ghosal S, Krzastek S, Rapp D, Ortiz N, Smith R. Is low-intensity shockwave therapy for erectile dysfunction a durable treatment option?-long-term outcomes of a randomized sham-controlled trial. Transl Androl Urol. 2024 Oct 31;13(10):2194-2200. doi: 10.21037/tau-24-329. Epub 2024 Oct 28. PMID 39507860
- [Derived] Kennady EH, Bryk DJ, Ali MM, Ratcliffe SJ, Mallawaarachchi IV, Ostad BJ, Beano HM, Ballantyne CC, Krzastek SC, Clements MB, Gray ML, Rapp DE, Ortiz NM, Smith RP. Low-intensity shockwave therapy improves baseline erectile function: a randomized sham-controlled crossover trial. Sex Med. 2023 Nov 11;11(5):qfad053. doi: 10.1093/sexmed/qfad053. eCollection 2023 Oct. PMID 37965376